CLINICAL TRIAL: NCT06959056
Title: Evaluating the Impact of Cryo-analgesia on Recovery After Double Lung Transplantation: a Pilot Study
Brief Title: Evaluating the Impact of Cryo-analgesia on Recovery After Double Lung Transplantation
Acronym: CRyoLTRiX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Hans Van Veer, MD, Consultant Thoracic Surgeon, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S68933; U1111-1320-5059 (Other: WHO)
Record Dates: First submitted 2025-03-31; First posted 2025-05-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Lung Transplant; Pain
Keywords: cryo nerve block; lung transplantation; cryoanalgesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryo nerve block + routine pain care (Active Comparator): Participants will undergo cryo nerve block at 6 levels of intercostal muscles, on each side from T3 to T8, 3cm lateral to the parasympathetic chain. The intervention will be performed after receptor pneumonectomy on each side.
  Interventions: Device: cryo nerve block at T3-T8 intercostal nerves bilaterally
- Routine pain care (No Intervention): Participants in the control arm will receive standard institutional pain care following bilateral lungtransplantation.

INTERVENTIONS:
Device: cryo nerve block at T3-T8 intercostal nerves bilaterally — In order to obtain better analgesia at the level of the chest wall, where the chest is bilaterally opened for lung extraction and donor lung implantation, intraoperative cryo-ablation will be applied to the intercostal nerves at the bilateral intercostal spaces 3-8, 3cm lateral to the sympathetic chain, under direct visualization during surgery, as such covering 2 intercostal levels above as well as below the normal access of ICR 4 or 5. By providing analgesia to level 8, we will also cover the area of chest drains, which also tend to cause pain in the postoperative course, especially when patients start mobilizing at the ward. Each nerve bundle will be cooled to a temperature between -65 and -72 °C during 120 seconds by means of the CyroSphere v2 probe (AtriCure Inc; Mason, OH, USA) connected to the provided instrument tower (AtriCure CryoICE box) including a processor device measuring and regulating the N2O flow through the probe.
  Arms: Cryo nerve block + routine pain care

SUMMARY:
The goal of this pilot trial is to learn whether the use of cryo nerve block and its effect on sensation in the chest alters recovery after bilateral lung transplantation, and to which extent these parameters are influenced. As this study is setup as a pilot study, the main questions it aims to determine the potential impacted parameters as well as their effect sizes, of cryo-analgesia on both short and long term outcomes following bilateral lung transplantation in COPD patients in a European high volume lung transplant centre.

The efficacy parameters under evaluation will be:

* is the highest pain score affected by the use of cryo nerve block?
* Is there an effect on the lung function ?
* Does cryo nerve block cause specific complications?
* are patients treated with cryo nerve block still needing the same amount of morphine as a pain killer?
* is the length of stay in intensive care influenced by the use of cryo nerve block?
* and is the qualiy of life influenced by the use of cryo nerve block?

Participants will:

* undergo cryo nerve block or receive routine pain treatment after bilateral lung transplantation
* be followed up during the first week after the operation, and every month to determine their pain
* be asked to perform a lung function test and complete quality of life questionnaires 1, 2, 3, 6 months and 1 year after transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. At least 18 years of age at the time of signing the Informed Consent Form (ICF)
3. Bilateral lung transplantation at UZ Leuven
4. Indication for transplantation: End stage chronic obstructive pulmonary disease (COPD)
5. Storage of lungs on classic ice, cooled system (LUNGguard® (Paragonix) or X°Port Lung Transport Device (Traferox Technologies Inc.) ) are all permitted
6. Patients that have undergone lung volume reduction or talcage are not a contraindication for participation in the study.

Exclusion Criteria:

1. Unilateral lung transplantation
2. Lobar transplantation
3. Donor lung reconditioning using ex-vivo lung perfusion (EVLP)
4. Combined organ transplantation
5. Chronic opioid use pre-operatively
6. Participation in an interventional Trial with an investigational medicinal product (IMP) or device (IMD) that could potentially influence the post-operative outcomes of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue pain Scale value | Postoperative days 0 to 7, 14, and 21 and every month postoperative until 1 year postoperative
  The highest pain score throughout the day in a participant, expressed on a Visual Analogue Scale instrument for assessing pain will be recorded. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Lung function | 1, 2, 3, 6 and 12 months postoperative
  Lung function evaluated by spirometry, recorded as Forced Expiratory Value at one second and Functional Vital Capacity expressed in liters and percentage of the expected.
opioid consumption | postoperative days 1-7, and every monthly contact until 1 year postoperative
  use of iv or oral morphin derivatives including tramadol, as well as transdermal delivery forms, expressed in oral morphine milligram equivalents (OMME)
Length of stay (LOS) at ICU | from transplantation until actual discharge of the intensive care unit, between 2 days and 6 months postoperative
  length of stay at the intensive care unit, expressed in days
Total hospital length of stay (HLOS) | from treatment until last day in the hospital of the index admission, between 2 days and 6 months postoperative
  total length of hospital stay, expressed in days
Evaluation of Quality of life - SF12 | single time points at 1, 2, 3, 6 months and 1 year postoperative
  Evaluation of quality of life by completion of standardized Quality of Life questionnaire (Short Form -12 (SF12)); 5 point likert scale; higher score equals better quality of life
Evaluation of Quality of life - EQ5D5L | single time points at 1, 2, 3, 6 months and 1 year postoperative
  Evaluation of quality of life by completion of standardized Quality of Life questionnaire (Evaluation of Quality of Life in 5 domains at 5 levels (EQ5D5L)); minimum score 5, maximum score 25; lower score equals better quality of life
Evaluation of Quality of life - Brief Pain Inventory | single time points at 1, 2, 3, 6 months and 1 year postoperative
  Evaluation of quality of life by completion of standardized Quality of Life questionnaire (Brief Pain Inventory); lower score equals better quality of life
Evaluation of Neuropathic Pain | single time points at 1, 2, 3, 6 months and 1 year postoperative
  Evaluation of pain characteristics in order to probe for neuropathic pain levels by means of the Neuropathic Pain Assessment questionnaire; 5 point likert scale, higher score is worse

CONTACTS AND LOCATIONS:
Overall Officials: Hans Van Veer, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Laurens Ceulemans, MD, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven; Yanina Jansen, MD, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
Data embargo imposed by the research institution